CLINICAL TRIAL: NCT01907971
Title: Left Ventricular Function in Ebstein Anomaly: Assessment by 3D Echocardiography and Speckle Tracking. Assessment and Validation of the Right Ventricle by VentriPoint Method.
Brief Title: Assessment of Left and Right Ventricular Function in Patients With Ebstein Anomaly With Different Echocardiographic Methods
Status: Completed | Type: Observational
Sponsor: Angela Oxenius (Other)
Collaborators: University Hospital, Zürich (Other)
Responsible Party: Sponsor-Investigator, Angela Oxenius, MD, University Children's Hospital, Zurich
Organization: University Children's Hospital, Zurich (Other)
Other Study IDs: VentriPoint in Ebstein anomaly
Record Dates: First submitted 2013-07-22; First posted 2013-07-25 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2014-03

CONDITIONS: Ebstein Anomaly
MeSH Terms: conditions — Ebstein Anomaly

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Ebstein anomaly: Patients with Ebstein anomaly

SUMMARY:
Ebstein anomaly is a rare congenital heart disease. It encompasses abnormalities of the tricuspid valve, the right atrium and the right ventricle (RV).

Currently, cardiac magnetic resonance imaging (MRI) is considered the method of choice for the assessment of RV volume and function. To evaluate the right heart function VentriPoint method was designed to assess the RV in a fraction of the time, resulting in better efficacy and lower costs. VentriPoint is approved for Tetralogy of Fallot patients as well as patients with systemic RV in d-transposition of the great arteries. This method uses 2 dimensional standard ultrasound views linked to a VentriPoint Medical Systems unit. After acquisition, the physician identifies anatomical landmarks with dots on a number of the 2D ultrasound views through the heart. With a sensor (magnetic tracking system: GPS) on the ultrasound probe we know where the 2D plane is in 3D space. In this way the precise anatomical landmark is located in 3D space.

The aim of the present study is to assess the feasibility, reliability and accuracy of the echocardiographic knowledge-based 3D reconstruction method to measure RV volume and function in patients with Ebstein anomaly. The accuracy of the method will be assessed by comparison with measurements obtained by cardiac MRI.

In addition to the right ventricle the investigators want to assess the left ventricular function in patients with Ebstein anomaly in this study. By using speckle tracking echocardiography the investigators would like to investigate on the left ventricular contractility, rotation and synchrony of the left ventricle together with the RV. Not seldom the left ventricle is neglected in a patient with Ebstein anomaly by impressive findings of the right ventricle. Changes in the myocardial left ventricular structure (non compaction) are also described and may have negative impact on the function.

The investigators want to analyze 25-30 patients with Ebstein anomaly including children starting at 11 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Ebstein anomaly
* male and female 11 years to 80 years of age
* Unoperated or operated on the heart, including 1 1/2 chamber palliation
* Wolff-Parkinson-White Syndrome

Exclusion Criteria:

* moderate or severe mitral valve insufficiency, moderate or severe aortic insufficiency, moderate or severe aortic stenosis
* Univentricular palliation (Fontan)
* St.n. myectomy of the left ventricle
* Concomitant L-transposition of the great arteries

Ages: 11 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Ebstein anomaly patients of the Zurich Area followed by primary care center
Sampling Method: Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2013-08; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Right ventricular volume (ml/m2) and function by VentriPoint. Structural myocardial changes in the left ventricle (Strain). | 1 year
  Comparison of the VentriPoint findings with measurements obtained by cardiac MRI.
  Structural changes of the left ventricle by echocardiography as well as ventricular longitudinal deformation in strain value by speckle tracking echocardiography.

SECONDARY OUTCOMES:
Correlation of findings with clinical symptoms | 1 year
  Correlation with the severity of tricuspid regurgitation, the clinical symptoms, size and function of the right ventricle

CONTACTS AND LOCATIONS:
Overall Officials: Christine H Attenhofer, Prof, Principal Investigator
Locations (1):
- University Childrens Hospital, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- See also: Related Info — http://www.ventripoint.com